CLINICAL TRIAL: NCT06550687
Title: Study of Cancer Patients' Preferences for Genetic Information Modalities Preceding Theranostic Exome Analysis. Qualitative Observational and Interventional Cross-sectional Study
Brief Title: Study of Cancer Patients' Preferences for Genetic Information Modalities Preceding Theranostic Exome Analysis.
Acronym: INFOGENE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 2024-A00091-46
Record Dates: First submitted 2024-08-06; First posted 2024-08-13 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: All Types of Metastatic Solid Malignancy; 1st-line Treatment; Exome Analysis; Active File EXOMA2 Study

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase 1:Observe communication between physicians and cancer patients (Other): * Observation of the 10 consultations : To ensure heterogeneous sampling, a varied panel of prescribing physicians will be selected, taking into account gender, age and specialty (oncologist versus organ specialist).
  * Conduct a semi-structured interview within 10 days of the consultation with 10 new patients who have been prescribed a theranostic exome analysis by a researcher
  * Thematic content analysis of 10 consultation observations by SHS researchers and 10 semi-structured interviews which will enable us to assess the degree of understanding of the information provided by the doctor, and whether it answers the patient's questions.
  Interventions: Other: Cancer patients' preferences regarding genetic information modalities prior to theranostic exome analysis
- Phase 2 : Revisit existing information media (GGC information note and video). (No Intervention): These materials will serve as a basis for our work, and may be adapted according to the results of phase 1 of our study. We will seek the advice of a partner patient, who will himself have benefited from a genetic analysis in the context of cancer, and who will be made aware of clinical research.
- Phase 3:Assess patients' preferences with regard to 3 information modalities (Other): * A medical consultation, during which the doctor will provide each of the 60 patients with the standard form of information, together with the explanatory note (INFOGene study)
  * Within 10 days, a semi-structured interview with 30 of the 60 patients. These 30 patients will be selected to ensure maximum socio-demographic and clinical (cancer location) heterogeneity.
  * Division of the 60 patients into 3 groups of 20 stratified according to age, gender and cancer location, including 10 previously interviewed (one group will receive the information based solely on the video worked previously, one group will receive the information during a consultation, one group will receive the information first via the video and then during a consultation).
  * The researcher conducts a new semi-structured interview with the 60 patients. They will provide an insight into patients' experience of the information they receive (content, form, timing).
  Interventions: Other: Cancer patients' preferences regarding genetic information modalities prior to theranostic exome analysis

INTERVENTIONS:
Other: Cancer patients' preferences regarding genetic information modalities prior to theranostic exome analysis — Phase 1: Observation of doctor-patient consultations Phase 2: Adaptation of information tools Phase 3: Assessment of understanding of information tools
  Arms: Phase 1:Observe communication between physicians and cancer patients; Phase 3:Assess patients' preferences with regard to 3 information modalities

SUMMARY:
Currently, the EXOMA2 study (NCT04614480) offers earlier and more comprehensive exome analysis in the management of cancer patients than EXOMA. Based on the active EXOMA2 patient file, the INFOGene study offers the opportunity to study patient-physician communication, to assess patient preferences with regard to different information modalities concerning theranostic exome analysis, and to reflect on information modalities to ensure optimal patient comprehension of the information provided.

The qualitative cross-sectional study includes a dual observational and interventional component involving cancer patients. The patients will come from the EXOMA 2 active file at Dijon University Hospital and the CGFL.

DETAILED DESCRIPTION:
Currently, the EXOMA2 study (NCT04614480) offers earlier and more comprehensive exome analysis in the management of cancer patients than EXOMA. Based on the active EXOMA2 patient file, the INFOGene study offers the opportunity to study patient-physician communication, to assess patient preferences with regard to different information modalities concerning theranostic exome analysis, and to reflect on information modalities to ensure optimal patient comprehension of the information provided.

The qualitative cross-sectional study includes a dual observational and interventional component involving cancer patients. The patients will come from the EXOMA 2 active file at Dijon University Hospital and the CGFL.

Phase 1 will aim to observe and analyze interpersonal communication between physicians prescribing theranostic exome analysis and cancer patients. It will be based on:

1/ ethnographic exploratory observations of 10 consultations during which the doctor will suggest that the patient undergo theranostic exome analysis, and 2/ semi-directed interviews with 10 new patients who have previously seen the doctor.

The patients will come from the EXOMA 2 active file at Dijon University Hospital and the CGFL.

* Step 1a : - construction of a consultation observation grid (based on existing literature) / - identification and inclusion of patients and physicians observed
* Step 1b : Observation of 10 consultations with a varied panel of prescribing physicians, taking into account taking into account gender, age, specialty and a heterogeneous sample of patients in socio-demographic and clinical terms
* Step 1c : semi-structured interview within 10 days of the consultation with consultation with 10 other patients by an SHS researcher to assess the degree of of the information provided by the doctor and whether it can be used to respond to the patient's needs.
* Step 1d : thematic content analysis

Phase 2 will consist in revisiting existing information supp orts (genetic counselor's explanatory note and and video). These materials will serve as a basis for work, and can be adapted according to the needs of the client.

Phase 3 will aim to evaluate patients' preferences with respect to 3 information modalities concerning a theranostic exome analysis.

* Step 3a: medical consultation, during which the doctor will provide each of the 60 patients with the standard form of information reworked by the in phase 2
* Step 3b : semi-structured interview within 10 days with researcher with 30 of the 60 patients.
* Step 3c : 60 patients divided into 3 groups of 20 stratified by age, gender and cancer site.

and cancer location, including 10 seen in interview:

* one group will receive information based solely on the video previously previously
* one group will receive information during a consultation
* one group will receive information first via the video and then during a consultation
* Step 3d : A new semi-structured interview with the 60 patients. These interviews will be carried out within 2 weeks of the information phase, in order to limit memory bias but also to allow time for the patients to express themselves.

ELIGIBILITY:
Inclusion Criteria:

* Patient identified for inclusion in the EXOMA 2 study (exome analysis request)
* Available to receive different types of information
* Fluent in French
* No prior oncogenetic consultation
* Having been informed of the objectives of the study and having given written non-objection to participate in the INFOGene study
* Authorizing audio recording of consultations and interviews

Exclusion Criteria:

* Patient who refused to participate in the EXOMA2 study (for phase 3 patients only)
* Has a psychiatric, cognitive or neurological disorder that makes participation impossible
* Working in the field of genetics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-09-19 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Concepts of communication and preferences. | Through study completion, an average of 21 months.
  The various interviews (phases 1 and 3) will provide an insight into patients' level of health literacy, which may explain the ease or difficulty of exchanges with the doctor (phase 1), as well as patients' preferences for one type of information over another (phase 3).

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre Georges-François Leclerc, Dijon
  - CHU François Mitterand, Dijon

IPD SHARING:
Plan to Share IPD: No